CLINICAL TRIAL: NCT06866912
Title: Observational Epidemiological Study of Patients Suffering From Systemic Amyloidosis
Acronym: AMI-ER
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: AMI-ER
Record Dates: First submitted 2025-01-29; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: Cardiomyopathy
Keywords: Cardiac amyloidosis
MeSH Terms: conditions — Cardiomyopathies; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
observational epidemiological study of patients affected by systemic amyloidosis

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with amyloidosis or asymptomatic carriers of mutations in the transthyretin gene
* minimum age of 18 years at the time of diagnosis
* obtaining informed consent

Exclusion Criteria:

* nothing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all adult patients referred to the participating centers with a diagnosis of amyloidosis or carriers of pathogenic mutations starting from 01/01/1981 diagnosed in accordance with current international guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2033-08-31 (Estimated); Study Completion 2033-08-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of amyloidosis | throughout the study period until 10 years
  prevalence of amyloidosis in patients admitted to the UOs participating in the study
incidence of amyloidosis | throughout the study period until 10 years
  incidence of amyloidosis in patients admitted to the UOs participating in the study
Observational epidemiological study of patients with systemic amyloidosis | throughout the study period until 10 years
  characteristics of each etiology in terms of baseline clinical data
Types of cardiac clinical phenotype | throughout the study period until 10 years
  Cardiac clinical phenotype in patients who at baseline are asymptomatic carriers of pathogenic mutations
Incidence of mixed clinical phenotype | throughout the study period until 10 years
  Mixed clinical phenotype in patients who at baseline are asymptomatic carriers of pathogenic mutations
Incidence of hospitalization for heart failure | throughout the study period until 10 years
  Incidence during follow-up of hospitalization for heart failure
Incidence of hospitalization for onset of arrhythmias | throughout the study period until 10 years
  Incidence during follow-up of hospitalization for onset of arrhythmias
Incidence of hospitalization for stroke | throughout the study period until 10 years
  Incidence of hospitalization for stroke during follow-up
incidence of pacemaker implantation | throughout the study period until 10 years
  incidence during follow-up of need for pacemaker implantation
incidence of pacemaker implantation of defibrillator | throughout the study period until 10 years
  incidence during follow-up of need for defibrillator implantation
Incidence of cardiac transplantation | throughout the study period until 10 years
  incidence during follow-up of need for cardiac transplantation
Incidence of transplantation of other solid organs | throughout the study period until 10 years
  incidence during follow-up of need for other solid organ transplantation
Mortality | throughout the study period until 10 years
  total mortality during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Simone Longhi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
Confidenciality